CLINICAL TRIAL: NCT02591303
Title: Stress and Insomnia: Investigating a Bidirectional Relation
Brief Title: Stress and Insomnia
Acronym: StresSleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Labex Brain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2015/12
Record Dates: First submitted 2015-10-16; First posted 2015-10-29 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Insomnia; Stress
Keywords: Insomnia; Stress; Real-life stressful events
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insomnia group (Experimental): Patients with insomnia: sleep complaints, of more than 3 nights a week, more than 3 months, affected daytime functioning, objectified low sleep quality (Sleep Efficiency <85%) with 10 days actigraphy
  Interventions: Other: Stress reactions measurement during stressful and neutral driving sessions
- Control group (Experimental): No sleep problems either self reported or objectified through actigraphy (Sleep Efficiency >85%)
  Interventions: Other: Stress reactions measurement during stressful and neutral driving sessions

INTERVENTIONS:
Other: Stress reactions measurement during stressful and neutral driving sessions — Stress effects will be measured during 3 driving sessions (training without events on Day 17, with neutral events on Day 18, with stressful events on Day19), through nighttime PSG and questionnaires.

SUMMARY:
Insomnia is characterized by rumination and worry over stressful events affecting nighttime sleep. Emotional reactions while stressful events are ongoing have not often been investigated in insomnia. In the current study stress reactions will be measured during a real-life simulation experiment with stressful events and investigate not only how previous sleep patterns affect emotional reactivity to the event but also how the emotional events affect sleep patterns the following night.

Thirty-six female subjects (age 25-45 years) without sleep complaints (n=18) or with insomnia (n=18) will enroll in a interventional study measuring the reaction to and effects of either neutral or stressful events during driving. Through questionaires and intake polysomnography, clinical levels of depression and anxiety will be excluded as well as sleep medication use and alternative sleep disorders than insomnia. Stress levels will be measured through skin conductance and heart rate variability during events and through nighttime polysomnography (PSG). Effects on sleep architecture and arousal levels will be measured through nighttime PSG.

Investigators hypothesize that subjects with insomnia, compared to subjects without sleep complaints, show stronger emotional reactions to stressful events and stronger effects of stress on sleep quality the following night. Results will facilitate a model for emotional reactivity in chronic sleep disruption which may aid to prevent short term sleep disruption converting into chronic insomnia and aid in developing customized insomnia treatment.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia group: patients with insomnia (DSM-V criteria): sleep complaints, of more than 3 nights a week, more than 3 months, affected daytime functioning
* Control group: no self-reported sleep problems
* 20-50 years old
* Female
* Having given written informed consent to participate in the research project
* Driving license

Exclusion Criteria:

* Night and shift-workers,
* Psychiatric disorder: clinical mood disorder, anxiety disorder, psychosis, bipolar disorder,
* For insomnia group: all sleep disorders other than persistent insomnia,
* For control group: all sleep disorders
* Progressive neurological diseases that include restless legs syndrome,
* Cardiovascular disease other than treated hypertension,
* Unstable respiratory or endocrinological diseases,
* Reporting symptoms of menopause and/or taking hormone replacement therapy for menopause symptoms,
* Drug addiction, alcohol addiction during the previous 6 months (smoking is allowed),
* Having undertaken trans-meridian travel (± 3H) in the previous 1 month,
* Pregnant or lactating women.
* Chronic pain.
* Having simulator-sickness during the first practice session
* Hypnotic and psychotropic medication taking or stopped less than 5 half-life periods of molecules before screening V0.
* A change in skin conductance of less than 0.05 microSiemens after an auditory stimulus.
* Left-handedness
* Patient participating to any other interventional study

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

PRIMARY OUTCOMES:
Heart rate variability at the stressful event | Day 19 after pre-inclusion
Skin conductance changes at the stressful event | Day 19 after pre-inclusion
  Electrodermal responsiveness is defined as a change in skin conductance with a minimum amplitude of 0.05 microSiemens
Reaction times at the stressful event | Day 19 after pre-inclusion

SECONDARY OUTCOMES:
Total sleep time by polysomnography | Days 17, 18 and 19 after pre-inclusion
Rapid Eye Movement (REM) duration by polysomnography | Days 17, 18 and 19 after pre-inclusion
Non-Rapid Eye Movement (NREM) duration by polysomnography | Days 17, 18 and 19 after pre-inclusion
Sleep spindle density by polysomnography | Days 17, 18 and 19 after pre-inclusion
Total sleep time obtained by actimetry | Every night between pre-inclusion and Day 20 (study termination)
Sleep efficiency obtained by actimetry | Every night between pre-inclusion and Day 20 (study termination)
Wake after sleep onset obtained by actimetry | Every night between pre-inclusion and Day 20 (study termination)
Sleep latency obtained by actimetry | Every night between pre-inclusion and Day 20 (study termination)
Visual analogue scale for driving stressfulness | Days 17, 18 and 19 after pre-inclusion
Presleep State Arousal Scale | Days 10, 18, 19 and 20 after pre-inclusion
PostTraumatic Stress Disorder checklist | Day 20

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France